CLINICAL TRIAL: NCT02330185
Title: Phase IV Study of Landmarks for Spinal Anesthesia
Brief Title: Comparison of Two Anatomic Landmarks With Ultrasonography in Spinal Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, İBRAHİM ÖZTÜRK, Phase IV Study of Landmarks for Spinal Anesthesia, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Screening
Other Study IDs: SALANDMARKUSG
Record Dates: First submitted 2014-11-06; First posted 2015-01-01 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Arthropathy of Knee
Keywords: spinal anesthesia; ultrasonography; anatomical landmark
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- spinal anesthesia for knee arthroscopy (Experimental): The intervention is spinal anesthesia. Tenth rib line or Tuffier's line will be examined as application landmarks by ultrasonography for spinal anesthesia.
  Interventions: Device: ultrasonography

INTERVENTIONS:
Device: ultrasonography — spinal anesthesia guided with ultrasonography

SUMMARY:
The most used anatomical landmark for application of spinal anesthesia is Tuffier's line. Other alternative landmark is tenth rib. However there is no trial that compare these landmarks based on using ultrasonography.

DETAILED DESCRIPTION:
The investigators aim to compare two landmarks (Tuffier's line and tenth rib line) for accuracy by using ultrasonography. 40 patients will be included in each groups. all of them will be assessed by ultrasonography during application of spinal anesthesia. And the investigators will examine the percentage of successful estimation of correct vertebral space.

ELIGIBILITY:
Inclusion Criteria:

* knee arthroscopic surgery

Exclusion Criteria:

* BMI>30
* anatomical anomaly of vertebrae

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2015-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
success of estimation the correct vertebral space | 2 months
  Independently, first anesthesist will determine the spinal anesthesia application point (intervertebral space) according to Tuffier's line and second anesthesist will determine it by ultrasonography. And third anesthesist will compare the accuracy of first determination.

CONTACTS AND LOCATIONS:
Overall Officials: dilek yazıcıoğlu, Study Chair — anesthesiology and reanimation

REFERENCES:
- [Background] Jung CW, Bahk JH, Lee JH, Lim YJ. The tenth rib line as a new landmark of the lumbar vertebral level during spinal block. Anaesthesia. 2004 Apr;59(4):359-63. doi: 10.1111/j.1365-2044.2004.03657.x. PMID 15023107